CLINICAL TRIAL: NCT04255953
Title: Development of a Telehealth Obesity Intervention for Patients With MS: Modifying Diet and Exercise in MS
Acronym: MoDEMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jared Bruce (Other)
Collaborators: National Multiple Sclerosis Society (Other); University of Kansas Medical Center (Other); Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor-Investigator, Jared Bruce, Professor, Biomedical & Health Informatics, University of Missouri, Kansas City
Organization: University of Missouri, Kansas City (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 2016418; RG-1901-33239IRB (Other Grant/Funding Number: MS Society)
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis; Obesity
MeSH Terms: conditions — Multiple Sclerosis; Obesity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (Active Comparator): Following baseline assessment, patients randomized to the TAU arm will receive monthly dietary pamphlets and web-based obesity prevention educational materials from the U.S. Office of Disease Prevention and Health Promotion (https://healthfinder.gov/HealthTopics/). After the 6-month assessment, TAU patients will begin the weight loss intervention arm.
  Interventions: Behavioral: behavioral telehealth; Other: Treatment as Usual
- Group Telehealth Obesity (Experimental): Participants will receive 24 weekly group phone counseling sessions and monthly individual sessions that encourage healthy eating and exercise. The planned intervention is guided by a social-cognitive framework and includes self-monitoring, goal setting, stimulus control, social support, cognitive reframing of unrealistic and negative thoughts, and developing positive expectancies for long-term weight control. The primary objective is to decrease caloric intake and increase physical activity to produce weight loss of approximately .4 to.9 kg per week, with the study goal of 10% reduction from baseline.
  Interventions: Behavioral: behavioral telehealth

INTERVENTIONS:
Behavioral: behavioral telehealth — Participants will receive 24 weekly group phone counseling sessions. Each session will last approximately 60 minutes and begin with an open-ended check-in question, followed by review of weekly self-monitoring data, question and answer time, and end with a new didactic topic of the week addressing diet, physical activity, or behavior change topics. Participants will be instructed to follow a diet that is reduced to 1200-1500 kcal/day and includes ≥ 5 fruit and vegetable (FV) servings per day, <25% kcal from fat, and 20-30 g of fiber. Physical activity will be gradually increased through a guided home-based program. Throughout the intervention, self-monitoring will be emphasized as a key behavioral weight loss strategy.
Other: Treatment as Usual — Treatment as Usual
  Arms: Treatment as Usual

SUMMARY:
We will tailor a telehealth obesity intervention for obese patients with MS (figure 2). Half of the patients will be randomly assigned to 24 weekly hour-long group weight loss sessions and 6 monthly individual sessions; half will be assigned to a brief education/Treatment as Usual (TAU) control condition. Participants assigned to the control condition will also receive the active treatment 6 months following their enrollment. As such, we will have feasibility, acceptability, and outcome data for all patients who enroll and complete the intervention. During outpatient recruitment, clinicians will ask obese patients (WHtR >.57, BMI >29) if they would be willing to be contacted about a study investigating a weight loss intervention for patients with MS. Patients who express interest and respond to advertisements will be screened by telephone and via review of medical records. Patients who meet initial eligibility criteria will be invited for a baseline evaluation where they will be formally consented, complete questionnaires and behavioral tasks, and undergo a standardized physical exam. They will be monitored using actigraphy for 10 days. They will then be randomized to the group telehealth obesity intervention or TAU. At 6 months, all participants will undergo a second in-person follow-up assessment and TAU participants will begin the telehealth intervention. At 12 months, participants will undergo a third in-person assessment, providing treatment outcome data for all study participants and long-term weight maintenance data for patients initially assigned to the telehealth obesity intervention. At 18 months, participants initially assigned to the TAU control condition will undergo a 4th assessment, providing weight maintenance data for all enrolled participants.

ELIGIBILITY:
Inclusion Criteria:

(a) a diagnosis of relapsing-remitting, secondary progressive, or primary progressive MS based on established guidelines and verified by medical chart review (b) between the ages of 18-70 (c) access to a telephone (d) English-speaking (e) ability to walk 25 feet without assistance and no severe sensory or motor impairment that would limit participation or present serious medical risks (f) no medically confirmed relapse in the past month (g) no history of dementia or severe cognitive difficulties that would limit participation (h) WHtR >.57 or BMI >29 (i) no history of bariatric surgery (j) no history of food allergies or need for a special diet preventing consumption of the recommended diet (k) no concurrent ongoing behavioral or pharmacological weight loss interventions (l) no history of insulin dependent diabetes or serious pulmonary/cardiac conditions (m) weight stability with no history of >10 pounds weight loss or gain in the 3 months prior to study participation (n) no planned or recent joint replacement surgeries (o) no serious psychiatric disorder (e.g. schizophrenia), current suicidal ideation, or current binge eating disorder as these patients may not be good candidates for behavioral weight loss programs (p) no current medical conditions where weight loss is contraindicated, as indicated by the participant's primary care physician (q) no contraindications to exercise (answer "no" to all 7 questions on Physical Activity Readiness Questionnaire; PAR-Q114) or physician approval to exercise if answer "yes" to 1 or more questions on PAR-Q. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 6 months
  percent weight change

SECONDARY OUTCOMES:
modified fatigue Impact scale | 6 months
  self-reported fatigue
Hospital Anxiety and Depression Scale | 6 months
  self-reported depression
MS Quality of Life Inventory | 6 months
  Self-report measure of quality of life
6 Minute Walk | 6 months
  Mobility Assessment

OTHER OUTCOMES:
Actigraphy | 6 Months
  Change in Activity pre/post treatment
DXA | 6 Months
  Body composition/Percent body fat

CONTACTS AND LOCATIONS:
Overall Officials: Jared Bruce, PhD, Principal Investigator — University of Missouri, Kansas City
Locations (1):
- University of Missouri-Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No